CLINICAL TRIAL: NCT00005450
Title: Health Promotion in the Elderly--Prevention of Cardiovascular Disorders
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4380; R43HL044280 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Cerebrovascular Disorders
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Cerebrovascular Disorders

SUMMARY:
To develop an epidemiologic model to estimate the benefits, costs and risks of disease prevention in the elderly.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

The investigators extended work they had done in modeling the health benefit of reducing risk factors for cardiovascular disease. Their new model incorporating risks of importance in the elderly, including cerebrovascular disease, estimated both morbidity and mortality averted by risk reduction, and estimated the costs and risks of the interventions used to modify risk factors.

The model was designed for the counseling of elderly individuals free of cardiovascular disease, and evaluated strategies for remaining disease free. It was implemented as software running on personal computers, and marketed to physicians and other health professionals who advised the elderly on medical issues. Accompanying documentation was also developed to explain the assumptions and non-quantifiable aspects of the decision to adopt major lifestyle changes to reduce risk.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-05; Study Completion 1991-11 (Actual)